CLINICAL TRIAL: NCT03177174
Title: the General Hospital of PLA
Brief Title: Different Chemotherapy Protocols Combined With Intensity Modulated Radiation Therapy in Patients With Locally Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luo yanrong (Other)
Responsible Party: Sponsor-Investigator, Luo yanrong, Clinical Doctor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2017-030-02
Record Dates: First submitted 2017-03-18; First posted 2017-06-06 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
Keywords: locally advanced nasopharyngeal carcinoma; Concurrent chemoradiotherapy; Toxic reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Cisplatin (Active Comparator)
  Interventions: Drug: Cisplatin
- DocetaxelCisplatin (Active Comparator): Cisplatin combined with Docetaxel
  Interventions: Drug: Cisplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Cisplatin — radiotherapy combined with Chemotherapy Drugs, Cancer
  Arms: Cisplatin; DocetaxelCisplatin
Drug: Docetaxel — Docetaxel
  Arms: Docetaxel; DocetaxelCisplatin

SUMMARY:
This study was to evaluate the efficacy ,toxic reaction and safety of different chemotherapy combined with radiotherapy on patients with locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18, <70 years old, with locally advanced nasopharyngeal carcinoma.

Exclusion Criteria:

* patients who had accepted radiotherapy before patients with any ather types of cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
changes in toxic reaction | 5 years
  incidence rate of the toxic reaction between three groups

SECONDARY OUTCOMES:
over survival | 5 years
  differences of over survival rate between three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA general hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Y, Cai B, Li B, Liu F, Du L, Zhao D, Fan W, Meng L, Zhang X, Ma L. The Acute Toxicities and Efficacy of Concurrent Chemotherapy With Docetaxel Plus Cisplatin, or Docetaxel, or Cisplatin and Helical Tomotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma: A Randomized Single-Center Phase II Trial. Technol Cancer Res Treat. 2022 Jan-Dec;21:15330338221109974. doi: 10.1177/15330338221109974. PMID 35770295